CLINICAL TRIAL: NCT01815645
Title: Evaluating the Efficacy of Including Contingency Management to Standard Ambulatory Treatment for Crack Addiction - A Randomized Controlled Trial
Brief Title: Contingency Management Treatment for Crack Addiction - Study With Brazilian Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, André de Queiroz Constantino Miguel, Ph.D Studant, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/01469-7 (FAPESP)
Record Dates: First submitted 2013-03-18; First posted 2013-03-21 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Cocaine Related Disorders
Keywords: Cocaine related disorders; Contingency Management; psychosocial treatment
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Masking Description: Both participants and researchers know the treatment alocations
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment Alone (Active Comparator): Participants in the Standard Treatment Alone group will receive 12 weeks of the exact treatment provided by the Ambulatory service where the study is being conducted
  Interventions: Behavioral: standard treatment
- ST+CM (Experimental): Participants in the Standard treatment plus Contingency Management (ST+CM) group will receive 12 weeks of the exact treatment provided by the Ambulatory service where the study is being conducted plus CM.
  Interventions: Behavioral: ST+CM

INTERVENTIONS:
Behavioral: ST+CM — 12 weeks of the standard treatment offered by a open treatment service for drug addiction of the city of Sao Paulo (AME) plus Contingency Management
  Arms: ST+CM
Behavioral: standard treatment — 12 weeks of standard treatment offered by AME (a open treatment service for drug addiction of the city of Sao Paulo)
  Arms: Standard treatment Alone

SUMMARY:
Crack addiction has become a severe health problem in Brazil. Today, crack addiction is the primary cause for inpatient treatment for all illicit substances. When compared to cocaine, crack users develop much faster diagnoses for crack dependence, shows a more compulsive pattern of use, has higher probability of living or have lived in the streets, and of engaging in illegal activities. Consequently to this, mortality of crack addicts is 7 times higher than for the rest of the population.

Despite all efforts being made for the development of effective pharmacological treatments for stimulant addiction (crack included), up to today, there is no robust evidence of efficacy of any pharmacological treatment. For that reason, the use of evidence based psychosocial interventions is so important for treating this population.

Although today open treatment facilities in Brazil are more and more starting to use evidence-based interventions such as motivational interviewing, cognitive behavior therapy, relapse prevention and coping skills, such treatments present very modest results when treating crack addiction. The biggest difficulties encountered when treating this population are maintaining patients in treatment, reducing crack use and achieving continued abstinence.

A psychosocial treatment based in behavioral principals' named Contingency Management (CM) is widely applied in the USA. Recent meta-analyses and review studies present robust evidence that, when applied alone or in adjunction with other psychosocial and pharmacological treatment, CM is the most effective treatment for what regards, treatment retention, reducing drug use and promoting continued abstinence.

The purpose of this study is to evaluate if Contingence Management (CM) can be affective in the treatment of crack addiction in Brazil. To accomplish this, 60 individuals (male and female from 18 to 65 years of age) seeking open treatment for crack addiction will be randomized to 2 treatment conditions (Standard treatment (ST) or ST+CM. Both treatments will last 12 weeks with 3 and 6-month follow-up. In both groups patients will be encourage to leave urine samples 3 times week.

Hypotheses: Patients receiving ST+CM will stay longer in treatment, have more negative tests for cocaine/crack, and achieve longer periods of cocaine/crack abstinence when compared to patients receiving ST alone.

DETAILED DESCRIPTION:
This study is a Randomized Clinical Trial deigned to investigate the effects of including Contingency Management to a standard public ambulatory treatment in Brazil on treatment attendance, retention in treatment, reduction of crack cocaine use and promotion of crack cocaine abstinence for crack dependent individuals seeking treatment for there addiction. In total 65 subjects will be randomized to receive Standard Treatment Alone or Standard Treatment plus Contingency Management. Both interventions will last for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnose of crack addiction (DSM IV)
* having used crack in the last month

Exclusion Criteria:

* Current psychotic disorder
* Diagnose of schizophrenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronaldo R Laranjeira, PhD, Principal Investigator — EPM/UNIFESP
Locations (1):
- Ambulatorio Medico de Especialidades (AME) da Vila Maria, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miguel AQ, Madruga CS, Cogo-Moreira H, Yamauchi R, Simoes V, da Silva CJ, McPherson S, Roll JM, Laranjeira RR. Contingency management is effective in promoting abstinence and retention in treatment among crack cocaine users in Brazil: A randomized controlled trial. Psychol Addict Behav. 2016 Aug;30(5):536-543. doi: 10.1037/adb0000192. Epub 2016 Jul 21. PMID 27442691
- [Derived] de Queiroz Constantino Miguel A, Sandi Madruga C, Simoes V, Yamauchi R, da Silva CJ, McDonell M, McPherson S, Roll J, Laranjeira RR, de Jesus Mari J. Contingency management is effective in promoting abstinence and retention in treatment among crack cocaine users with a previous history of poor treatment response: a crossover trial. Psicol Reflex Crit. 2019 Jul 15;32(1):14. doi: 10.1186/s41155-019-0127-2. PMID 32026092
- [Derived] Miguel AQC, Madruga CS, Cogo-Moreira H, Yamauchi R, Simoes V, Ribeiro A, da Silva CJ, Fruci A, McDonell M, McPherson S, Roll JM, Laranjeira RR. Contingency management targeting abstinence is effective in reducing depressive and anxiety symptoms among crack cocaine-dependent individuals. Exp Clin Psychopharmacol. 2017 Dec;25(6):466-472. doi: 10.1037/pha0000147. PMID 29251975

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Treatment: standard treatment: 32 participants received 12 weeks of standard treatment offered by AME (a open treatment service for drug addiction of the city of Sao Paulo)
- Standard Treatment Plus Contingency Management: 33 participants received Standard treatment plus Contingence Management: 12 weeks of the standard treatment offered by a open treatment service for drug addiction of the city of Sao Paulo (AME) plus Contingency Management
Period: Overall Study
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management
Started | 32 | 33
Completed | 32 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Treatment Plus Contingency Management: Standard treatment plus Contingence Management: 12 weeks of the standard treatment offered by a open treatment service for drug addiction of the city of Sao Paulo (AME) plus Contingency Management
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 33 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (8.5) | 35.3 (8.7) | 35.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 26 | 30 | 56
Region of Enrollment [Number; unit: participants]
  Brazil | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Longest Duaration of Achieved Abstinance
Description: Number of Participants with 4, 8 and 12 Weeks Continued Abstinence
Time Frame: 12 weeks of treatment
Population: Longest duaration of abstinance was determined by the highest amount of consecutive negative crack/cocaine samples submitted.
Measure: Number; unit: number of participants
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management
Number analyzed (Participants) | 32 | 33
number of participants
  12 weeks of abstinance | 0 | 7
  8 weeks of abstinance | 1 | 8
  4 weeks of abstinance | 1 | 12

2. Primary Outcome: Percentage Samples Submitted Negative for Crack Cocaine Use
Description: Proportion of samples testing negative for Crack Cocaine use
Time Frame: 12 weeks
Measure: Number; unit: percentage of submitted negative samples
Units Other Than Participants: urine samples
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management
Number analyzed (Participants) | 32 | 33
Number analyzed (urine samples) | 113 | 628
percentage of submitted negative samples | 8.3 | 46.5

3. Primary Outcome: Number of Participants Completing 4, 8 and 12 Weeks of Treatment
Description: Retention in treatment was quantified as the period elapsed between treatment intake and dropout (last appearance at the treatment facility) or the end of treatment. We present data on the number of participants retained in treatment in weeks 4, 8 and 12.
Time Frame: Number of participant retained in treatment at weeks 4, 8 and 12.
Measure: Number; unit: number of participants
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management
Number analyzed (Participants) | 32 | 33
number of participants
  Retained in week 12 | 0 | 17
  Retained in week 8 | 8 | 21
  Retained in week 4 | 11 | 22

4. Primary Outcome: Treatment Attendance
Description: Treatment attendance was expressed as the total number of sessions attended during the 12 weeks of treatment.
Time Frame: 12 weeks
Population: we compared group means for the total number of attended sessions.
Measure: Mean (Standard Deviation); unit: attended treatment sessions
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management
Number analyzed (Participants) | 32 | 33
attended treatment sessions | 3.7 (5.9) | 19.5 (14.9)

5. Secondary Outcome: Percentage Samples Submitted Negative for Alcohol Use
Description: Proportion of samples testing negative for alcohol use
Time Frame: 12 weeks
Measure: Number; unit: percent of sample
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management
Number analyzed (Participants) | 32 | 33
percent of sample | 9.4 | 53.9

6. Secondary Outcome: Percentage Samples Submitted Negative for Marihuana Use
Description: The proportion of samples testing negative for marijuana was determined by dividing the number of negative samples by the total number of expected samples (36 samples)
Time Frame: 12 weeks
Measure: Number; unit: percent of sample
Units Other Than Participants: percent of sample
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management
Number analyzed (Participants) | 32 | 33
Number analyzed (percent of sample) | 36 | 36
percent of sample | 9.8 | 50.3

ADVERSE EVENTS:
Arm/Group | Standard Treatment | Standard Treatment Plus Contingency Management
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 0/32 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No